CLINICAL TRIAL: NCT03682939
Title: Evaluation of Safety and Immunogenicity of Meningococcal B and Meningococcal ACWY Vaccine in at Risk Population (ProPositive Study)
Brief Title: Evaluation of Safety and Immunogenicity of Meningococcal B and Meningococcal ACWY Vaccine in at Risk Population
Acronym: ProPositive
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17.0177
Record Dates: First submitted 2018-09-13; First posted 2018-09-25 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Hiv; Meningitis, Meningococcal; HIV Infections
Keywords: vaccination; HIV; meningitis; Vaccine; Immunogenicity; Safety; Bexsero; Menveo; co-administration
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Meningitis, Meningococcal; HIV Infections; Meningitis | interventions — 4CMenB vaccine; Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Single arm, open-label, all participants will receive both Bexsero® (meningitis B vaccine) and Menveo® (meningitis ACWY vaccine) vaccines.
  Interventions: Biological: Bexsero® (meningitis B vaccine); Biological: Menveo® (meningitis ACWY vaccine)

INTERVENTIONS:
Biological: Bexsero® (meningitis B vaccine) — Bexsero® 0.5ml IM vaccine administered into non-dominant arm of participant
Biological: Menveo® (meningitis ACWY vaccine) — Menveo® 0.5ml IM vaccine administered into dominant arm of participant

SUMMARY:
This study aims to evaluate the immunogenicity, safety and tolerability of co-administration of vaccinations for meningitis B (Bexsero®) and meningitis ACWY (Menveo®) in adults and children aged 10-45 years living with HIV. All participants will be vaccinated with both Menveo® and Bexsero® on days 0 and 30. Immunogenicity will be determined on venous blood sampled at days 0 and 60. Adverse effects will be recorded to evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

* Any 10-45-year old male or female patients with confirmed HIV infection where they (or someone with parental responsibility) can sign fully informed consent and are able to comply with study requirements.

Exclusion Criteria:

* Pregnancy or breast feeding,
* History of MenACWY (Menveo® or Nimenrix®) and 4CMenB (Bexsero®) vaccination in the previous 2 years,
* Receipt of other non-live vaccines within 2 weeks and live vaccines within 4 weeks of first dose, planned receipt of vaccine within 2 weeks of study visits,
* Current active malignancy,
* Known latex allergy
* Known or suspected hypersensitivity to any components of the vaccines or history of severe allergic reaction after previous vaccination
* Bleeding disorder preventing IM vaccination,
* Any acute or chronic illness which according to the investigators judgement would prevent patients to receive the vaccines or participate in the study
* Participation in clinical trials concerning investigational medical product within 0 days or before completion of the study
* Children in care

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in hSBA geometric mean titres to relevant strains of meningococcal B following two doses of the 4CmenB vaccine (Bexsero®) in people living with HIV | Day 0 (baseline) and Day 60
  The human complement serum bactericidal assay (hSBA) mean titres against relevant strains of meningococcal B at baseline and one month after completion of vaccination.
The proportion of participants who achieve at least a four fold increase in hSBA titres. | Day 60
  Blood will be taken one month after the second vaccine and serum tested for hSBA titres. The proportion of participants who achieve at least a four fold increase in hSBA titres will be calculated.
The proportion of participants who achieve a 'protective' hSBA titre of >1:4 after two doses of Bexsero | Day 60
  Blood will be taken one month after the second vaccine and serum tested for hSBA titres. The proportion of participants who are deemed to have protective titres >1:4 will be calculated.

SECONDARY OUTCOMES:
The incidence of solicited and unsolicited adverse and serious adverse events after two doses of MenACWY (Menveo®) and 4CMenB (Bexsero®) vaccines when co-administered in people living with HIV | Day 7 after vaccines 1 and 2
  We will assess the following:
  1. The incidence of subjects with solicited local and systemic AEs up to 7 days (including the day of vaccination) after Visits 1 and 2.
  2. The incidence of subjects with any other (unsolicited) AEs, including any SAEs, AEs leading to withdrawal and medically attended AEs up to 7 days (including the day of vaccination) after Visits 1 and 2.
  3. The incidence of subjects with SAEs and AEs leading to withdrawal throughout the study period.
The geometric mean titres to Meningococcal ACWY antigens after two doses of the MenACWY (Menveo®) vaccine in people with HIV at one month after the second vaccination | Day 60
  We will measure rSBA GMTs for MenACWY antigens at baseline and Visit3.
The proportion of subjects with at least a four fold change in rSBA from baseline to 30 days after the second vaccine | Day 0 and Day 60
  The proportion of subjects with at least 4 fold increase in rSBA against relevant MenACWY serogroups from baseline to Visit3.
The proportion of subjects with "protective" rSBA titres >1:8 against relevant MenACWY serogroups after two doses of Menveo | Day 60
  The proportion of subjects with "protective" rSBA titres >1:8 against relevant MenACWY serogroups at Visit3.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cosgrove, MBBS PhD, Principal Investigator — St George's, University of London
Locations (1):
- St Georges University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simmons RD, Kirwan P, Beebeejaun K, Riordan A, Borrow R, Ramsay ME, Delpech V, Lattimore S, Ladhani S. Risk of invasive meningococcal disease in children and adults with HIV in England: a population-based cohort study. BMC Med. 2015 Dec 9;13:297. doi: 10.1186/s12916-015-0538-6. PMID 26654248
- [Background] Dwilow R, Fanella S. Invasive meningococcal disease in the 21st century-an update for the clinician. Curr Neurol Neurosci Rep. 2015 Mar;15(3):2. doi: 10.1007/s11910-015-0524-6. PMID 25637287
- [Background] Miller L, Arakaki L, Ramautar A, Bodach S, Braunstein SL, Kennedy J, Steiner-Sichel L, Ngai S, Shepard C, Weiss D. Elevated risk for invasive meningococcal disease among persons with HIV. Ann Intern Med. 2014 Jan 7;160(1):30-7. doi: 10.7326/0003-4819-160-1-201401070-00731. PMID 24166695
- [Background] Cohen C, Singh E, Wu HM, Martin S, de Gouveia L, Klugman KP, Meiring S, Govender N, von Gottberg A; Group for Enteric, Respiratory and Meningeal disease Surveillance in South Africa (GERMS-SA). Increased incidence of meningococcal disease in HIV-infected individuals associated with higher case-fatality ratios in South Africa. AIDS. 2010 Jun 1;24(9):1351-60. doi: 10.1097/QAD.0b013e32833a2520. PMID 20559040
- [Background] Cohn AC, MacNeil JR, Clark TA, Ortega-Sanchez IR, Briere EZ, Meissner HC, Baker CJ, Messonnier NE; Centers for Disease Control and Prevention (CDC). Prevention and control of meningococcal disease: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2013 Mar 22;62(RR-2):1-28. PMID 23515099
- [Background] Frota AC, Milagres LG, Harrison LH, Ferreira B, Menna Barreto D, Pereira GS, Cruz AC, Pereira-Manfro W, de Oliveira RH, Abreu TF, Hofer CB. Immunogenicity and safety of meningococcal C conjugate vaccine in children and adolescents infected and uninfected with HIV in Rio de Janeiro, Brazil. Pediatr Infect Dis J. 2015 May;34(5):e113-8. doi: 10.1097/INF.0000000000000630. PMID 25876102
- [Background] Lujan-Zilbermann J, Warshaw MG, Williams PL, Spector SA, Decker MD, Abzug MJ, Heckman B, Manzella A, Kabat B, Jean-Philippe P, Nachman S, Siberry GK; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1065 Protocol Team. Immunogenicity and safety of 1 vs 2 doses of quadrivalent meningococcal conjugate vaccine in youth infected with human immunodeficiency virus. J Pediatr. 2012 Oct;161(4):676-81.e2. doi: 10.1016/j.jpeds.2012.04.005. Epub 2012 May 22. PMID 22622049
- [Background] Findlow J, Bai X, Findlow H, Newton E, Kaczmarski E, Miller E, Borrow R. Safety and immunogenicity of a four-component meningococcal group B vaccine (4CMenB) and a quadrivalent meningococcal group ACWY conjugate vaccine administered concomitantly in healthy laboratory workers. Vaccine. 2015 Jun 26;33(29):3322-30. doi: 10.1016/j.vaccine.2015.05.027. Epub 2015 May 27. PMID 26025807
- [Background] Santolaya ME, O'Ryan ML, Valenzuela MT, Prado V, Vergara R, Munoz A, Toneatto D, Grana G, Wang H, Clemens R, Dull PM; V72P10 Meningococcal B Adolescent Vaccine Study group. Immunogenicity and tolerability of a multicomponent meningococcal serogroup B (4CMenB) vaccine in healthy adolescents in Chile: a phase 2b/3 randomised, observer-blind, placebo-controlled study. Lancet. 2012 Feb 18;379(9816):617-24. doi: 10.1016/S0140-6736(11)61713-3. Epub 2012 Jan 18. PMID 22260988
- [Derived] Isitt C, Bartolf A, Andrews N, Athaide S, Pryce-Williams R, Townsend-Payne K, Borrow R, Ladhani S, Heath PT, Cosgrove CA. The propositive study: Immunogenicity and safety of a four-component recombinant protein-based vaccine against MenB and a quadrivalent conjugate MenACWY vaccine in people living with HIV. HIV Med. 2023 Sep;24(9):979-989. doi: 10.1111/hiv.13495. Epub 2023 Apr 23. PMID 37088964